CLINICAL TRIAL: NCT03167281
Title: Early Intrapleural TPA Instillation Versus Late
Acronym: ELEVATE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of adequate recruitment
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00058518
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Tissue Plasminogen Activator
Keywords: Chest tube; Thoracostomy; Pleural Diseases; Lung Neoplasms; Pulmonary Embolism; Pneumothorax; Thoracic Surgery; Deoxyribonucleases; Fibrinolytic Agents; Drainage; Pleural Effusion
MeSH Terms: conditions — Pleural Diseases; Lung Neoplasms; Pulmonary Embolism; Pneumothorax; Pleural Effusion | interventions — Deoxyribonucleases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- tPA and DNase (No Intervention): 10mg of t-PA and 5 mg of DNase in a 30 mL solution of water/saline administered via chest tube over three days twice daily 24-48 hours after chest tube placed.
- Early tPA and DNase (Experimental): 10mg of t-PA and 5 mg of DNase in a 30 mL solution of water/saline administered via chest tube over three days twice daily with initial administration occurring at chest tube placement.
  Interventions: Combination Product: early tPA and DNase

INTERVENTIONS:
Combination Product: early tPA and DNase — Early addition of tPA and DNase (immediately at chest tube placement) versus later (24-48 hours) after chest tube placement.
  Arms: Early tPA and DNase

SUMMARY:
Chest tubes are used for air or fluid removal from the pleural space. When a chest tube is placed, it can be hard for the fluid to drain.Tissue plasminogen activator (tPA) and DNase are given through the chest tube to help with draining the fluid. We are doing this research to see if early addition of tPA-DNase immediately after chest tube placement will help with better fluid draining.

DETAILED DESCRIPTION:
The purpose of this study is to determine the timing and efficacy of early administration and late administration of t-PA/DNase via thoracostomy (n=60). Patients will be identified from the Intensive Care Unit, Coronary Care Unit, and wards/stepdown units. Prior to chest tube placement, patients will be randomized to one of the two treatment arms (early use of t-PA-DNase verus late use of t-PA-DNase). Route of administration will be via their thoracostomy tube over a period of three days twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18 years or older
* Patients with an indication for a thoracostomy tube placement for a pleural effusion

Exclusion Criteria:

* Patients that require a thoracostomy tube for a pneumothorax
* Pregnant women
* Sensitivity to t-PA, or DNase
* Patients taking carbamazepine or nitroglycerin
* Lung volume reduction surgery on side of pleural effusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Chest tube removal | 7 days
  Time to chest tube removal

SECONDARY OUTCOMES:
Fluid drainage | 3 days
  Volume of fluid drained after each tPA and DNase instillation
Need for other interventions | 4 days
  Post tPA/DNase administration, the need for other interventions, such as surgery or additional chest tube, will be determined.
Discharge | 3 weeks
  Time to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Mankikar, MD, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Palmetto Health Richland, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: South Carolina Research Studies Directory — http://scresearch.org/studies/search?utf8=%E2%9C%93&q=Mankikar&commit=GO